CLINICAL TRIAL: NCT02294786
Title: A Randomised, Multicentre, Open Label, Phase II Study of Prophylactic Octreotide to Prevent or Reduce the Frequency and Severity of Diarrhoea in Subjects Receiving Lapatinib With Capecitabine for the Treatment of Metastatic Breast Cancer
Brief Title: Study of Prophylactic Octreotide to Prevent or Reduce the Frequency and Severity of Diarrhoea in Subjects Receiving Lapatinib With Capecitabine for the Treatment of Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117314
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Results first posted 2019-07-15 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: Randomised; Octreotide; Diarrhoea; Phase II; Capecitabine; Quality of life; Metastatic breast cancer; HER2; Lapatinib; Diarrhoea diary
MeSH Terms: conditions — Neoplasms; Diarrhea; Breast Neoplasms | interventions — Lapatinib; Capecitabine; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Octreotide treatment (Experimental): Subjects randomised to receive Octreotide were administered with Octreotide (Sandostatin LAR™) 40mg 7 days before the start of treatment with Lapatinib and Capecitabine and again 28 days later. All subjects received treatment with Lapatinib 1250milligram (mg) once daily and Capecitabine 1000 milligram/square meter (mg/m^2) twice daily until disease progression. Lapatinib was given every day; Capecitabine was given in 3 week cycles of two weeks treatment followed by one week off treatment. SANDOSTATIN™ is a trademark of Novartis.
  Interventions: Drug: Lapatinib; Drug: Capecitabine; Drug: Octreotide
- No Octreotide treatment (Experimental): Subjects randomised to receive no octreotide, treatment with Lapatinib and Capecitabine was initiated immediately following enrolment. All subjects received treatment with Lapatinib 1250mg once daily and Capecitabine 1000mg/m^2 twice daily until disease progression. Lapatinib was given every day; Capecitabine was given in 3 week cycles of two weeks treatment followed by one week off treatment
  Interventions: Drug: Lapatinib; Drug: Capecitabine

INTERVENTIONS:
Drug: Lapatinib — Lapatinib was supplied as 250mg tablets that are oval, biconvex, and orange film-coated with one side plain and the opposite side debossed, or as 250mg tablets that are oval, biconvex, and yellow film-coated with one side plain and the opposite side debossed. Each tablet contained 405mg of Lapatinib ditosylate monohydrate, equivalent to 250mg Lapatinib free base
Drug: Capecitabine — Capecitabine (Xeloda™) was supplied as a biconvex, oblong, light peach or peach colored film-coated tablet for oral administration. Each light peach colored tablet contained 150mg Capecitabine and each peach colored tablet contained 500mg Capecitabine. Generic versions of capecitabine may have been used within the study if Xeloda cannot be provided. XELODA™ is a trademark of Hoffmann-La Roche AG.
Drug: Octreotide — Octreotide (Sandostatin LAR™) was supplied as sterile 5milliliter (mL) vials delivering 20mg Octreotide as the free peptide. When mixed with diluent (approximately 2mL or 2.5 mL) it becomes a suspension that is given as an intramuscular injection. Two 20mg intramuscular injections were given to deliver a total dose of 40mg. The Octreotide is uniformly distributed within the microspheres which are made of a biodegradable glucose star polymer, D,L-lactic and glycolic acids copolymer. Sterile mannitol was added to the microspheres to improve suspendability
  Arms: Octreotide treatment

SUMMARY:
Diarrhoea is the most commonly reported adverse event (AE) associated with Lapatinib treatment, and is also commonly associated with Capecitabine treatment. Although these events are generally mild to moderate in severity, diarrhoea adversely affects the tolerability of cancer treatment, and in severe cases diarrhoea has the potential to affect the efficacy of treatment due to poor compliance, or treatment interruption or withdrawal. The efficacy of Octreotide in the management of cancer treatment-associated diarrhoea has not been extensively evaluated in large, well-controlled studies. This is a randomised, multi-centre, open-label Phase II study in subjects with Human epidermal growth factor receptor 2 (HER2)-positive metastatic breast cancer which has progressed following prior therapy, which must have included anthracyclines and taxanes and therapy with Trastuzumab in the metastatic setting. This study is not placebo controlled, and there is no active comparator. The study evaluates whether the prophylactic use of Octreotide Long Acting Release (LAR) offers a clinically meaningful benefit by reducing the frequency and severity of diarrhoea associated with treatment with Lapatinib and Capecitabine. Study completion for a subject is defined as the completion of 24 weeks of treatment with Lapatinib and Capecitabine, or progression of cancer or the death of the subject during treatment, whichever occurs first. Approximately 140 subjects were planned to be randomized out of which 70 were planned to receive octreotide and 70 were planned to receive no Octreotide.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Histologically or cytologically confirmed HER2-positive advanced or metastatic breast cancer which has progressed following prior therapy, which must have included anthracyclines and taxanes and therapy with trastuzumab in the metastatic setting
* Females age >=18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy of at least 12 weeks
* Able to swallow and retain oral medications
* Incapable of becoming pregnant, or not pregnant and using an adequate form of contraception, i.e. a female who is of:

  1. non-childbearing potential (physiologically incapable of becoming pregnant), including any female who has had hysterectomy, bilateral oophorectomy, bilateral tubular ligation or is post-menopausal (total cessation of menses for at least 1 year);
  2. childbearing potential must have a negative serum pregnancy test within 7 days prior to treatment with Octreotide if randomised to receive Octreotide or the first dose of Lapatinib with Capecitabine if randomised to receive no Octreotide, preferably as close to the first dose as possible, and must agree to use adequate contraception (intrauterine device, birth control pills unless clinically contraindicated, or barrier device) and other acceptable contraceptive methods during the study and continuing for at least 4 weeks after the final dose of treatment with Lapatinib and Capecitabine
* Subjects must complete all screening assessments as outlined in the protocol
* Subjects must complete the Functional Assessment of Chronic Illness Therapy-Diarrhoea (FACIT-D) and diarrhoea diary before receiving the first dose of Octreotide if randomised to receive Octreotide. All subjects must complete the FACIT-D and diarrhoea diary before receiving the first dose of Lapatinib with Capecitabine
* Prior treatment with other chemotherapeutic agents or endocrine therapy is permitted. All prior treatment related toxicities, except diarrhoea and alopecia, must be National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) (version 4.03)<= Grade 1 at the time of randomization.Subjects with diarrhoea with any grade of severity within 14 days prior to randomisation are excluded from LAP117314
* Prior treatment with radiation therapy is permitted provided that at least 2 weeks have elapsed since the last fraction of radiation therapy prior to treatment with Octreotide if randomised to receive Octreotide or the first dose of Lapatinib with Capecitabine if randomised to receive no Octreotide, and all radiation therapy related AEs are <= Grade 1 at the time of randomization
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria:

* Concurrent treatment with an investigational agent or concurrent participation in another clinical study
* Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to treatment with Octreotide for subjects randomised to receive Octreotide or the first dose of Lapatinib and Capecitabine for subjects randomised to receive no Octreotide
* Treatment with Octreotide within the 3 months prior to randomization
* Concurrent chemotherapy, radiation therapy, immunotherapy, biologic therapy (including an Epidermal growth factor receptor (EGFR) and/or HER2 inhibitor), or hormonal therapy for treatment of cancer
* Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent, unless a legally acceptable representative could provide informed consent (if in accordance with the policies of the local Ethics Committee)
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical or psychiatric disorder that would interfere with the subject's safety or compliance with study procedures
* Diarrhoea with any grade of severity within 14 days prior to treatment with Octreotide for subjects randomised to receive Octreotide or within 14 days prior to the first dose of Lapatinib and Capecitabine for subjects randomised to receive no Octreotide
* Malabsorption syndrome, inflammatory bowel disease (ulcerative colitis, Chrohn's disease), irritable bowel syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel
* Pregnant or lactating subjects
* Prior treatment with Lapatinib
* French subjects: the French subject has participated in any study using an investigational drug during the previous 30 days or 5 half-lives, whichever is longer, preceding the first dose of protocol treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2017-10-19 (Actual); Study Completion 2017-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- Novartis Investigative Site, Olomouc, Czechia
- Novartis Investigative Site, Tel Aviv, Israel
- Poland (3):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Warsaw
- Russia (6):
  - Novartis Investigative Site, Khanty-Mansiysk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Obninsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tomsk
- United Kingdom (4):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Romford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 62 women in 17 centers; Czech Republic (1), Israel (1), Poland (3), the United Kingdom (4) Russian Federation (8)
Pre-assignment Details: The study was terminated early after 62 patients (out of 140 planned) were randomized as criteria for futility was met.
Period: Overall Study
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Started | 30 | 32
Safety Population (All randomized subjects who received at least one dose of study treatment.) | 29 (One subject randomized to Octreotide received only 0.1 mg dose.) | 33 (The subject was included in the No-Octreotide arm.)
ITT Population (All randomized subjects regardless of whether or not treatment was administered.) | 30 | 32
Completed | 19 | 18
Not Completed | 11 | 14
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 6 | 7
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide Treatment | No Octreotide Treatment | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (10.07) | 55.9 (9.08) | 56.6 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Experiencing Diarrhoea of Grade 2 and Above (up to 24 Weeks)
Description: Proportion of subjects experiencing at least one episode of diarrhoea with a severity of Grade 2 and above, as defined by the National Cancer Institute common terminology criteria for adverse events (NCI CTCAE) version 4.03, recorded as AEs in the Electronic case report form (eCRF)
Time Frame: Up to 24 weeks
Population: ITT - For cycle 1-3 analysis: Subjects that withdrew from the study on or prior to the Cycle 4 visit date were assumed to have experienced diarrhoea. For the cycle 1-8 analysis: Subjects who did not have diarrhea event prior to the End of Study/Withdrawal visit date were not assumed to have experienced diarrhoea.
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants
  Cyclce 1-3 (up to 9 weeks)with impuation | 7 | 9
  Cyclce 1-8 (up to 24 weeks)without imputation | 6 | 5
Statistical Analysis 1: Comparison: Octreotide Treatment vs No Octreotide Treatment; Cycle 1-3 (up to 9 weeks); Test type: Superiority; p = 0.775, Chi-squared; Difference in Percentages = -4.8, 95% CI 2-sided [-29.2 to 20.0]

2. Secondary Outcome: Proportion of Subjects Experiencing Diarrhoea of Grade 3 and Above (up to 24 Weeks)
Description: Proportion of subjects experiencing diarrhoea with a severity of Grade 3 and above, as defined by the NCI CTCAE, version 4.03 and recorded as AEs in the eCRF
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 2 | 0

3. Secondary Outcome: Proportion of Subjects Experiencing Diarrhoea of Any Grade of Severity (up to 24 Weeks)
Description: Proportion of subjects experiencing diarrhoea of any grade of severity as defined by the NCI CTCAE, version 4.03 and recorded as AEs in the eCRF
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 18 | 14

4. Secondary Outcome: Duration of Diarrhoea of Any Grade of Severity
Description: Duration of diarrhoea of any grade of severity, recorded as AEs in the eCRF
Time Frame: Up to 24 weeks
Population: ITT - including only patients for whom an AE of diarrhoea and its duration was reported
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 17 | 13
days | 8.7 (11.15) | 36.8 (48.59)

5. Secondary Outcome: Time to Onset of the First Episode of Diarrhoea of Any Grade of Severity
Description: Time to onset of the first episode of diarrhoea of any grade of severity, recorded as an AE in the eCRF. Subject are censored if there was no event. Median time and 95% confidence intervals were calculated using Kaplan-Meier estimates.
Time Frame: Up to 24 weeks
Population: ITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Days | NA [54.0 to NA] — The median time to onset of first episode of diarrhea from the start of therapy was not reached. | 170 [104 to NA] — There were not enough events to calculate the upper 95% CI.

6. Secondary Outcome: Proportion of Subjects Taking Anti-diarrhoeal Medication
Description: Proportion of subjects taking anti-diarrhoeal medication as recorded in the eCRF
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 7 | 11

7. Secondary Outcome: Proportion of Subjects Who Had Unscheduled Visits to Healthcare Professionals Due to Diarrhoea
Description: Proportion of subjects making diarrhoea related unscheduled visits to healthcare professionals as recorded in the eCRF
Time Frame: Up to 24 weeks
Population: ITT - The information to calculate the proportions was not captured in the database.
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Proportion of Subjects Requiring Dose Reduction in Lapatinib and Capecitabine
Description: Proportion of subjects requiring diarrhoea related Lapatinib and Capecitabine dose reduction as recorded in the eCRF
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants
  Subjects requiring dose reduction in Lapatinib | 1 | 0
  Subjects requiring dose reduction in Capecitabine | 1 | 2

9. Secondary Outcome: Proportion of Subjects Requiring Dose Delay in Lapatinib and Capecitabine
Description: Proportion of subjects requiring diarrhoea related Lapatinib and Capecitabine dose delay as recorded in the eCRF
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants
  Subjects requiring dose delay in Lapatinib | 2 | 2
  Subjects requiring dose delay in Capecitabine | 2 | 2

10. Secondary Outcome: Proportion of Subjects Requiring Treatment Withdrawal in Lapatinib and Capecitabine
Description: Proportion of subjects requiring diarrhoea related Lapatinib and Capecitabine treatment withdrawal as recorded in the eCRF
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants
  Requiring treatment withdrawal in Lapatinib | 0 | 0
  Requiring treatment withdrawal in Capecitabine | 0 | 0

11. Secondary Outcome: Proportion of Subjects Requiring Use of Diarrhoea-related Intravenous Fluids
Description: Proportion of subjects requiring use of diarrhoea-related intravenous fluids for rehydration as recorded in the eCRF
Time Frame: Up to 24 weeks
Population: ITT - The information to calculate the proportions was not captured in the database.
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Lapatinib and Capecitabine Tablets Dispensed and Returned
Description: Number of Lapatinib and Capecitabine tablets dispensed and returned as recorded in the eCRF
Time Frame: Up to 24 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
tablets
  Number of Lapatinib tablets dispensed | 1197.5 (403.12) | 1115.6 (495.9)
  Number of Lapatinib tablets returned | 477.1 (173.94) | 403.3 (238.47)
  Number of Capecitabine tablets dispensed | 1022.6 (473.44) | 1011.2 (532.06)
  Number of Capecitabine tablets returned | 186.1 (157.19) | 210 (196.64)

13. Secondary Outcome: Overall Response Rate (up to 24 Weeks)
Description: Overall response rate as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >=20% and >= 5mm increase in the sum of diameters of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants
  complete response (CR) | 0 | 2
  partial response (PR) | 6 | 4
  stable disease (SD) | 4 | 5
  Progressive Disease | 14 | 17
  Not Evaluable | 6 | 4

14. Secondary Outcome: Clinical Benefit Response (up to 24 Weeks)
Description: Clinical benefit response as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  Clinical Benefit Response rate (CBR) is defined as the percentage of subjects with a CR, PR or SD at week 24.
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 7 | 9

15. Secondary Outcome: Proportion of Subjects Reporting Changes in Bowel Movements From Baseline (Frequency and/or Consistency) as Recorded in the Diarrhoea Management Diary (DMD)
Description: All subjects completed the baseline DMD during the 3 days prior to randomisation, before any study-related treatment is administered. Subjects randomised to receive Octreotide completed a second baseline DMD before starting the first cycle of treatment with Lapatinib and Capecitabine. The baseline DMD comprised of 3 questions to record stool form and consistency. The DMD to be completed throughout the rest of the study comprised of 3 questions in the baseline DMD and a further 5 questions and 6 sub-questions to evaluate the consequences and management of diarrhoea.
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 23 | 29

16. Secondary Outcome: Time to the First Subject Reported Change in Frequency and/or Consistency of Bowel Movements From Baseline as Recorded in the DMD
Description: Event is defined as Subjects reporting change in frequency and/or consistency of bowel movements from baseline at least once in DMD. Subject are censored if there is no change in bowel movement frequency/consistency as compared to baseline. Median time and 95% confidence intervals were calculated using Kaplan-Meier estimates.
Time Frame: Up to 24 weeks
Population: ITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Days | 22.0 [16.0 to 57.0] | 8.0 [8.0 to 15.0]

17. Secondary Outcome: Proportion of Subjects Taking Anti-diarrhoeal Medication as Recorded in the DMD
Description: The proportion of subjects taking medication at least once as a result of diarrhoea are summarised
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 2 | 2

18. Secondary Outcome: Proportion of Subjects Making Dietary Changes Due to Diarrhoea as Recorded in the DMD
Description: The proportion of subjects making dietary changes to help with the diarrhoea are summarised
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 9 | 11

19. Secondary Outcome: Proportion of Subjects Contacting Other Non-hospital Healthcare Professionals to Discuss Diarrhoea as Recorded in the DMD
Description: The proportion of subjects contacting a health care professional other than the hospital doctors/nurses to discuss diarrhoea are summarised
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 4 | 3

20. Secondary Outcome: Proportion of Subjects Reporting Stopping Completely or Missing Doses of Anti-cancer Tablets Due to Diarrhoea as Recorded in the DMD
Description: The proportion of subjects reducing or completely stopping the number of anti-cancer tablets to help with diarrhoea are summarised
Time Frame: Up to 24 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Treatment | No Octreotide Treatment
Number analyzed (Participants) | 30 | 32
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Up to 28 weeks post randomization (from randomization until up to and including 4 weeks after the last dose of study treatment)
Groups:
- Octreotide Treatment: Octreotide+Lap+Cap
- No Octreotide Treatment: Lap+Cap
- All Patients: All Patients
Arm/Group | Octreotide Treatment | No Octreotide Treatment | All Patients
All-Cause Mortality (participants affected / at risk) | 1/29 | 0/33 | 1/62
Serious Adverse Events (participants affected / at risk) | 5/29 | 3/33 | 8/62
Other Adverse Events (participants affected / at risk) | 26/29 | 27/33 | 53/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide Treatment (N=29) | No Octreotide Treatment (N=33) | All Patients (N=62)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Vulvitis (Infections and infestations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Paraparesis (Nervous system disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octreotide Treatment (N=29) | No Octreotide Treatment (N=33) | All Patients (N=62)
Anaemia (Blood and lymphatic system disorders) | 1 | 6 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 17 | 15 | 32
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 3
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 4
Oral pain (Gastrointestinal disorders) | 0 | 2 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 4
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3
Asthenia (General disorders) | 2 | 7 | 9
Fatigue (General disorders) | 3 | 1 | 4
Oedema peripheral (General disorders) | 2 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 2 | 4
Lower respiratory tract infection (Infections and infestations) | 3 | 1 | 4
Oral candidiasis (Infections and infestations) | 2 | 0 | 2
Paronychia (Infections and infestations) | 2 | 2 | 4
Alanine aminotransferase increased (Investigations) | 4 | 2 | 6
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 5
Bilirubin conjugated increased (Investigations) | 2 | 0 | 2
Blood bilirubin increased (Investigations) | 4 | 3 | 7
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 13 | 11 | 24
Rash (Skin and subcutaneous tissue disorders) | 4 | 7 | 11
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Lymphoedema (Vascular disorders) | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-09-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT02294786/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT02294786/SAP_001.pdf